CLINICAL TRIAL: NCT07294209
Title: Efficacy and Safety of Low-Dose Tenecteplase for Acute Ischemic Stroke Treatment in Aging Patients: A Prospective, Multicenter, Randomized Controlled Study
Brief Title: Low-Dose Tenecteplase for Acute Ischemic Stroke Treatment in Aging Patients
Acronym: DATE-AGING
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Zhenhua Zhou, Professor, Southwest Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025IITDA10
Record Dates: First submitted 2025-11-21; First posted 2025-12-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke Patients

STUDY DESIGN:
Intervention Model Description: multicenter, prospective, randomized, open label, blinded-endpoint (PROBE)，Parallel controls，Non-inferiority
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Dose Tenecteplase (Experimental): 0.175mg/kg tenecteplase
  Interventions: Drug: low-dose tenecteplase intravenous thrombolysis
- Standard-Dose Tenecteplase (Active Comparator): 0.25mg/kg tenecteplase
  Interventions: Drug: standard-dose tenecteplase intravenous thrombolysis

INTERVENTIONS:
Drug: low-dose tenecteplase intravenous thrombolysis — Subjects will be randomized to low-dose group or standard-dose group in a 1:1 ratio. Patients in the low-dose group received tenecteplase (0.175 mg/kg) for intravenous thrombolysis. The upper dose limit is set to 17.5 mg/patient.
  Arms: Low-Dose Tenecteplase
Drug: standard-dose tenecteplase intravenous thrombolysis — Subjects will be randomized to low-dose group or standard-dose group in a 1:1 ratio. Patients in the standard-dose group received tenecteplase (0.25 mg/kg) for intravenous thrombolysis. The upper dose limit is set to 25 mg/patient.
  Arms: Standard-Dose Tenecteplase

SUMMARY:
The DATE-AGING study is a prospective, multicenter, randomized controlled trial investigating low-dose tenecteplase in elderly patients with acute ischemic stroke. Its primary objective is to evaluate the safety and efficacy of low-dose tenecteplase in elderly patients within 4.5 hours of acute ischemic stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years;
2. Diagnosis of ischaemic stroke with a measurable neurological deficit on National Institutes of Health Stroke Scale (NIHSS) (1≤ NIHSS ≤25); if NIHSS <4, patients have to be with at least a measurable deficit on motor power (upper or lower limbs ≥1);
3. Stroke symptoms should have been present for at least 30 minutes (min) without significant improvement prior to randomisation;
4. Thrombolytic therapy can be initiated within 4.5 Hour(s) (h) of Acute ischaemic stroke (AIS) onset;
5. Patients with premorbid modified Rankin Scale (mRS) 0 or 1;
6. Informed consent from the patient or surrogate.

Exclusion Criteria:

1. Imaging demonstrates multi-lobar infarction (hypodensity >1/3 cerebral hemisphere);
2. Acute bleeding diathesis or allergy to tenecteplase, including but not limited to

   * Known genetic predisposition to bleeding or significant bleeding disorder at present or within the past 6 Month(s) (m)
   * Administration of heparin within the previous 48 h and activated partial thromboplastin time (aPTT) exceeding the upper limit of normal for laboratory measurement
   * Current use of vitamin K based oral anticoagulants (e.g. warfarin) and a prolonged prothrombin time (International normalised Ratio (INR) > 1.7 or Prothrombin time (PT)>15 seconds (s)) or current use of novel oral anticoagulants (i.e. dabigitran, rivaroxiban, or apixiban) with prolongation of activated partial thromboplastin time (aPTT) and/or PT above the upper limit of the local laboratory reference range
   * Platelet count of below 100×10^9/ L
   * Any history of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
   * Recent traumatic external heart massage or recent puncture of a non-compressive blood-vessel (e.g. subclavian or jugular vein puncture) , within the past 10 days
   * Known history of suspected intracranial haemorrhage or suspected subarachnoid haemorrhage from aneurysm
   * Neoplasm with increased haemorrhagic risk
   * Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial aneurysm, or arterial/venous malformations
   * History of significant trauma or major surgery within the past 3 months.
   * Any known disorder associated with a significant increased risk of bleeding
3. Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/extradural hematoma, etc.);
4. Blood glucose <2.8 mmol/L or >22.22 mmol/L;
5. After active antihypertensive treatment, hypertension is still not under control: systolic blood pressure ≥180 mmHg, or diastolic blood pressure ≥100 mmHg;
6. Seizure at stroke onset;
7. Concurrent malignancy or severe systemic disease with an anticipated survival of less than 90 days;
8. Participation in other clinical trials within 3 months prior to screening;
9. Unsuitability or participation in this study as judged by the Investigator may result in subjects being exposed to greater risk.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 798 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Modified Rankin Scale (mRS) Score of 0 or 1 | At Day 90±7 days
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death).

SECONDARY OUTCOMES:
Percentage of participants with major neurological improvement (National Institutes of Health Stroke Scale (NIHSS) score of 0 or improvement of at least 4 points compared with baseline) | At 24 hours
  National Institutes of Health Stroke Scale (NIHSS) is a 11-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 6 grades with 0 as normal, and there is an allowance for untestable items.Total NIHSS score (0-42) = sum of 11 individual item scores, higher total scores meaning more severe deficits.
Percentage of Participants With Modified Rankin Scale (mRS) Score of 0-2 | At Day 90±7 days
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death).
Distribution of Modified Rankin Scale (mRS) | At Day 90±7 days
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death).
Percentage of Participants With Barthel Index Score ≥95 | up to 90 days
  The Barthel Index is an ordinal scale used to measure performance in activities of daily living (ADL). The Barthel Index consists of 10 items. The total score of the Barthel Index ranges from 0 to 100, and higher scores indicate better outcome.
EQ-5D-5L score | At Day 90±7 days
  Health-related quality of life (the score on the EuroQol Group 5-Dimension 5-Level [EQ-5D-5L] questionnaire, range, -0.39 to 1, with higher scores indicating better quality of life)
Percentage of Participants With Symptomatic Intracerebral Haemorrhage (sICH) | up to 36 hours
  sICH via criteria adapted from the European Cooperative Acute Stroke Study (ECASS III), defined as any apparent extravascular blood in the brain or within the cranium that is associated with clinical deterioration defined by an NIHSS score increase of four points or more from baseline.
All-cause mortality | up to 90 days
  All-cause mortality at 90 days
Percentage of Participants With Modified Rankin Scale (mRS) Score of 5 or 6 | At Day 90±7 days
  Modified Rankin Scale (mRS) is a standardized measure that describes the extent of disability after a stroke. The mRS is a single item scale. It increases from 0 (no symptoms at all) to 6 (death).

CONTACTS AND LOCATIONS:
Locations (46):
- China (46):
  - Southwest Hospital, Chongqing, China, Chongqing, Chongqing Municipality
  - Anshan Changda Hospital, Anshan
  - Anyang People's Hospital, Anyang
  - Huaxian People's Hospital of Henan, Anyang
  - Baoshan People's Hospital, Baoshan
  - People's Hospital of Zhijin County, Bijie
  - Bishan Hospital, Chongqing
  - Chongqing Emergency Medical Center, Chongqing
  - Chongqing University Fuling Hospital, Chongqing
  - Chongqing University Jiangjin Hospital, Chongqing
  - Chongqing University Three Gorges Hospital, Chongqing
  - Dianjiang People's Hospital OF Chongqing, Chongqing
  - People's Hospital Of Xiushan County, Chongqing
  - The People's Hospital of Dazu Chongqing, Chongqing
  - The People's Hospital of HeChuan, Chongqing, Chongqing
  - The People's Hospital of Rongchang Chongqing, Chongqing
  - The People's Hospital of Tongnan District Chongqing City, Chongqing
  - The Seventh People's Hospital of Chongqing, Chongqing
  - Tongliang Hospital, Chongqing
  - Yunyang County People's Hospital, Chongqing
  - Dali Bai Autonomous Prefecture People's Hospital, Dali
  - Dazhou Central Hospital, Dazhou
  - The People's Hospital of Zhongjiang, Deyang
  - Guang an People's Hospital, Guang’an
  - Guizhou Provincial People's Hospital, Guiyang
  - The Second People's Hospital of Guiyang（Guiyang Jinyang Hospital）, Guiyang
  - The First Affiliated Hospital of Harbin Medical University, Ha’erbin
  - Xunxian People's Hospital, Hebi
  - Heyuan People's Hospital, Heyuan
  - The People's Hospital Of Jianyang City, Jianyang
  - Laixi People's Hospital, Laixi
  - People's Hospital of Leshan, Leshan
  - Luoyang Mengjin People's Hospital, Luoyang
  - Nanbu People's Hospital, Nanchong
  - Puyang People's Hospital, Pujiang
  - The People's Hospital of Nan Le Xian, Pujiang
  - People's Hospital of Ningling County, Shangqiu
  - The First People's Hospital of Shangqiu, Shangqiu
  - The First People ' S Hospital of Shao Yang, Shaoyang
  - Wuhan Puren Hospital, Wuhan
  - Xiangyang NO.1 People's Hospital, Xiangyang
  - The second people's hospital of Yibin, Yibin
  - Zhumadian Central Hospital, Zhumadian
  - Zhuzhou Central Hospital, Zhuzhou
  - Zigong Third People's Hospital, Zigong
  - Ziyang Central Hospital, Ziyang

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR